CLINICAL TRIAL: NCT01699308
Title: Growth Hormone and Brain Functioning After Traumatic Brain Functioning
Brief Title: Growth Hormone and Brain Functioning After Traumatic Brain Injury
Acronym: GH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Joe Springer (Other)
Responsible Party: Sponsor-Investigator, Joe Springer, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pfizer/WS935852; 09.0874-F1V (Other: UK IRB)
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Growth Hormone; Neuroimaging
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Genotropin (Experimental): 10 persons with TBI and GHD will receive daily rhGH injections titrated to bring their GH levels into the normal range for one year. Treatment is initiated using Genotropin (rhGH) at an initial daily dose of 200mcg/day subcutaneously with a titration schedule calling for an increase in daily dosage by 200 mcg every two months until the target daily dose, 600 mcg/day, is achieved. The 10 GHD subjects will be assessed at baseline with EEG, fMRI and DTI and neuropsychological measures, again at 6 months, and a third time at 12 months.
  Interventions: Drug: Genotropin
- Control (No Intervention): 5 demographically-matched TBI with normal GH subjects will be assessed at baseline (with EEG, fMRI and DTI, and neuropsychological measures) and at 12 months.

INTERVENTIONS:
Drug: Genotropin
  Other Names: somatropin
  Arms: Genotropin

SUMMARY:
The current protocol aims to compare the brain-functioning (fMRI & EEG) and white matter structural integrity (DTI) of persons with mild to severe TBI with and without Growth Hormone deficiency during cognitive tasks; and to examine changes in cognitive and motor performance, EEG/fMRI and white matter integrity associated with growth hormone treatment for twelve months using an open-label design in persons with GH deficiency/insufficiency following mild to severe TBI. To meet this aim, we are in the process of screening 40 persons with mild to severe TBI, ages 18-55, who are at least six months post injury. After screening, 10 persons with TBI and GHD (Growth Hormone deficiency) will receive daily rhGH injections titrated to bring their GH levels into the normal range over the course of twelve months. Treatment will be initiated using rhGH (Genotropin). Subjects with TBI and GHD will be assessed at baseline, 6 months, and 12 months with EEG, fMRI and DTI, and neuropsychological measures. 5 persons with TBI who do not have GHD will be assessed at baseline and at 12 months with EEG, fMRI and DTI, and neuropsychological measures.

ELIGIBILITY:
Inclusion Criteria:

* Mild to Severe TBI
* At Least 6 Months Post Injury
* Ages 18-55

Exclusion Criteria:

* Patients Taking Anticoagulants, Anticonvulsants, Cyclosporine, Corticosteroids, and Sex Steroids
* History of Hepatitis B or C
* History of Symptomatic Coronary Disease or Congestive Heart Failure
* Pre-Existing Neurologic Disease such as Epilepsy, Alzheimer's Disease, Multiple Sclerosis, Brain Tumors, etc.
* Obesity (BMI > 30)
* Pregnant or Lactating Females
* Penetrating Traumatic Brain Injury
* Having a Pacemaker
* Diabetes and Diabetic Retinopathy
* Serious Psychiatric Conditions (e.g., Schizophrenia, Bipolar Disorder, Major Depressive Disorder, etc.)
* Patients with Language Problems such as Aphasia
* Any Sign of Neoplastic Activity
* Active Malignancies
* Three-Fold Elevation of Liver Function Tests (ALP, ALT, AST)
* Partially Deficient in Both Cortisol and Thyroid
* Fully Deficient in Either Cortisol and Thyroid
* Patients with Claustrophobia
* Metal in the Body that Cannot be Removed (especially in the head)
* Amputations on Upper Body Limbs

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2009-12-01 (Actual); Primary Completion 2014-04-01 (Actual); Study Completion 2014-04-01 (Actual)

PRIMARY OUTCOMES:
Change in brain function assessed by functional MRI | baseline and one year
  Participants will undergo functional MRI at baseline and one year later to determine brain function after treatment. Data will be presented as the change in brain function over time presented as mean +/- SEM.
Change in brain function assessed by electroencephalogram | baseline and one year
  Participants will undergo electroencephalograms at baseline and one year later to determine brain function after treatment. Data will be presented as the change in brain function over time presented as mean +/- SEM.
Change in white matter structural integrity | baseline and one year
  Participants will undergo routine MRI at baseline and one year later. Data will be presented as the change in brain function over time presented as mean +/- SEM.

CONTACTS AND LOCATIONS:
Overall Officials: J Springer, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No